CLINICAL TRIAL: NCT00194558
Title: Outcomes and Cost Consequences of Using an Internet Co-Management Module to Improve the Quality of Type 1 Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 04-3892-G-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Health Education; Information Technology; Disease Management; Internet; Patient Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Health Education

INTERVENTIONS:
Behavioral: Internet co-management module

SUMMARY:
The researchers will conduct a 12-month randomized controlled trial comparing usual care versus chronic disease management using the Internet among patients with type 1 diabetes receiving care in the Diabetes Care Center at the University of Washington.

DETAILED DESCRIPTION:
We will conduct a 12-month randomized controlled trial comparing usual care versus chronic disease management using the Internet among patients with type 1 diabetes on multiple daily injections with insulin glargine and rapid-acting analogs. Specifically, the objectives of the study are to:

1. Evaluate the difference in glycemic control (HbA1c) between intervention and control,
2. Evaluate the difference in resource utilization and costs of care between intervention and control, and
3. Evaluate the difference in satisfaction with care between intervention and control.

A total of 80-85 subjects will be recruited from patients receiving care in the Diabetes Care Center (DCC) at the University of Washington in Seattle. As part of a pretest-posttest experimental design, intervention-group subjects will be trained in the use of an existing diabetes disease-management module comprising six related Web sites that are accessed from home via links displayed within the University's "MyUW" Internet portal. These sites allow patients to:

1. View their entire electronic medical record including clinical reminders, the same record used by providers,
2. Upload blood glucose readings stored in a digital meter,
3. Manually enter medication, nutrition, and exercise data into an online daily diary,
4. Communicate with providers regarding treatment recommendations or other questions using a clinical e-mail service,
5. Obtain additional information from a traditional education site whose content and links were sanctioned by the Medical Director of the DCC, and
6. Employ a second education site to collaboratively generate action plans intended to enhance self-efficacy.

In addition to login and password protection, access to confidential information from home requires the use of secondary authentication (SecureID). All clinical and other data can be viewed by patients and providers in online trended displays that will be used by a nurse practitioner to review cases no less than weekly. As the control group, subjects receiving usual care will not have access to the diabetes module and related case-management services being evaluated.

The primary clinical outcome for the study is the between group differences in glycemic control using HbA1c as the metric. A co-primary outcome is all direct medical care utilization. Satisfaction with diabetes care, employing both a quantitative survey (Patient Assessment of Chronic Illness Care) and semi-structured interviews performed on a 20% purposive sub-sample of intervention patients, is a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Computer and Internet access at home
* Receiving care at the University of Washington Diabetes Care Center

Exclusion Criteria:

* Non-English speaking

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2005-02

PRIMARY OUTCOMES:
Hemoglobin A1c

SECONDARY OUTCOMES:
Utilization
Satisfaction with care

CONTACTS AND LOCATIONS:
Overall Officials: Harold I Goldberg, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Diabetes Care Center, Seattle, Washington, United States